CLINICAL TRIAL: NCT03257436
Title: Strategic Management to Improve CRT Using Multi-Site Pacing Post Approval Study (Reference # C1918)
Acronym: SMARTMSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 92050975
Record Dates: First submitted 2017-08-18; First posted 2017-08-22 (Actual); Results first posted 2022-01-03 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Left Ventricular Dysfunction
Keywords: Pacing
MeSH Terms: conditions — Ventricular Dysfunction, Left

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Single Arm (Other): General population who receive a Boston Scientific Resonate family of CRT-D device in accordance with its labeled indication for use.
  Interventions: Device: CRT-D

INTERVENTIONS:
Device: CRT-D — Left Ventricular MultiSite Pacing

SUMMARY:
Prospective, multi-center, single arm, post approval study to be conducted in the United States.

DETAILED DESCRIPTION:
Evaluate the effectiveness of Boston Scientific (BSC)'s LV MSP (Left Ventricular MultiSite Pacing) feature in the Resonate family of CRT-D devices and confirm safety in a post approval study when used in accordance with its approved labeling.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who received de novo implantation of BSC's Resonate family of CRT-D devices with the LV MSP feature4 and BSC's ACUITYTM X4 LV Quadripolar leads. A Resonate family of CRT-D device upgrade from previous single or dual chamber pacemaker or ICD implantation is allowed.
2. Subjects must meet BSC labeled indication for CRT-D implantation.
3. Subjects must have a functional RA lead and RV lead implanted
4. Subjects who are willing and capable of providing informed consent
5. Subjects who are willing and capable of participating in all testing/visits associated with this clinical study at an approved clinical study center and at the intervals defined by this protocol
6. Subjects who are age 18 and above, or of legal age to give informed consent specific to state and national law

Exclusion Criteria:

1. Subjects who received LV pacing prior to receiving the Resonate family of CRT-D system implantation.
2. Subjects who received the LV MSP therapy post CRT-D implantation but prior to enrollment
3. Subjects with documented history of permanent AF
4. Subjects with documented permanent complete AV block
5. Subjects who are expected to receive a heart transplant during the 12 months course of the study
6. Subjects with documented life expectancy of less than 12 months
7. Subjects who enrolled in any other concurrent study or registry, with the exception of mandatory national or governmental registry, without prior written approval from BSC

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 586 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2020-11-19 (Actual); Study Completion 2020-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saba Samir, Principal Investigator — University of Pittsburgh Medical Center
Locations (54):
- United States (54):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Phoenix Cardiovascular Group, Phoenix, Arizona
  - Cardiology Associates of NEA, Jonesboro, Arkansas
  - Foothill Cardiology Medical Group, Arcadia, California
  - Chula Vista Cardiac Center, Chula Vista, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Desert Heart Rhythm Consultants, Palm Springs, California
  - Cardiology Associates Medical Group, Ventura, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Delray Medical Center, Delray Beach, Florida
  - UF Health Jacksonville, Jacksonville, Florida
  - Florida Hospital Waterman, Lake Mary, Florida
  - Tallahassee Research Institute, Tallahassee, Florida
  - Augusta University, Augusta, Georgia
  - Alexian Brothers Hospital Network, Elk Grove Village, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - Parkview Hospital Inc, Fort Wayne, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Norton Heart Specialist, Louisville, Kentucky
  - Advanced Cardiovascular Specialists, Shreveport, Louisiana
  - MedStar Heart and Vascular Institute, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Ascension St. John Hospital & Medical Center, Detroit, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - St. Mary's of Michigan Research Institute at Covenant Medical Ceter, Saginaw, Michigan
  - UMMC- Division of Cardiology, Jackson, Mississippi
  - St. Lukes Hospital, Kansas City, Missouri
  - Billings Clinic, Billings, Montana
  - Methodist Physicians Clinic Heart Consultants, Omaha, Nebraska
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Hackensack University Medical Canter, Hackensack, New Jersey
  - Montefiore Medical Center, The Bronx, New York
  - Durham VA medical Center, Durham, North Carolina
  - WakeMed, Raleigh, North Carolina
  - Trihealth- Good Samaritan & Bethesda North Hospitals, Cincinnati, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - St. Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Salem Health, Salem, Oregon
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Pinnacle Health Cardiovascular Institute, Wormleysburg, Pennsylvania
  - Berk Cardiologists, Wyomissing, Pennsylvania
  - AnMed Health Clinical Research, Anderson, South Carolina
  - Rapid City Regional Health, Rapid City, South Dakota
  - Stern Cardiovascular Foundation, Germantown, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Heartplace, PA, Bedford, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - UT Health, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Carient Heart and Vascular, Manassas, Virginia
  - Sentara Norfolk General, Norfolk, Virginia
  - St. Mary's Medical Center, Huntington, West Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm
Started | 584
Completed | 489
Not Completed | 95
Not completed — Withdrawal by Subject | 76
Not completed — Death | 19

BASELINE CHARACTERISTICS:
Population: Total subjects with non-missing values
Arm/Group | Single Arm
Number analyzed (Participants) | 583
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.7 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 211
  Male | 372
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 95
  White | 460
  More than one race | 10
  Unknown or Not Reported | 14
Region of Enrollment [Number; unit: participants]
  United States | 583

OUTCOME MEASURES:

1. Primary Outcome: LV MSP Feature Related Complication-Free Rate
Description: Proportion of subjects free from LVMSP feature related complications at 12 months
Time Frame: Between 6 month visit and the 12 month visit in non-responders with LV MSP on for any duration.
Population: Subjects who are non-responders at the 6 month follow up and who have LVMSP enabled for for any duration between the 6th and 12 month visit
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single Arm
Number analyzed (Participants) | 102
percentage of participants | 99 [94.1 to NA] — As prespecified in the study protocol the lower one-sided 95% confidence bound of the Kaplan-Meier estimate was compared to the performance goal (i.e., only the lower one-side confidence bound was necessary/utilized for hypothesis testing).
Statistical Analysis 1: Comparison: Single Arm; The LV MSP feature-related CFR between the 6 Month Visit and the 12 Month Visit was calculated using Kaplan-Meier methodology. H0: LV MSP feature-related complication-free rate between 6 Month Visit and 12 Month Visit ≤ 90%. The sample size of 61 subjects was required to evaluate the Primary Safety Endpoint using an exact test since a power calculation cannot be directly calculated for a one group Kaplan-Meier analysis; Test type: Other — A power calculation using a sample size of 61 subjects as the non-responders with the LV MSP on was calculated based on a one-sided exact test for a single binomial proportion, using SAS Version 9.4 with the following assumptions: * Performance goal = 90% * Expected LV MSP feature-related CFR rate between 6 and 12 Month Visit = 98% * Significance level = 5% * Power = 80%; Kaplan Meir Methodology = 99, 95% CI 1-sided [lower limit 94.1]

2. Primary Outcome: Proportion of LV MSP Group Subjects With an Improved Clinical Composite Score at 12 Months
Description: Proportion of non-responders with LV MSP enabled at 6 months who were responders at 12 months. Responders were defined as having an Improved Clinical Composite Score at 12 Months.
Time Frame: 12 Month Follow Up
Population: Non-responders at 6 Months who had LV MSP enabled and had complete clinical composite score data, LV MSP on and achieved >93% LVa and LVb pacing
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single Arm
Number analyzed (Participants) | 78
percentage of participants | 51.3 [41.4 to NA] — The 95% one-sided lower pointwise confidence limit of the response rate was calculated using the one-sided exact methodology for a single binomial proportion and compared to the performance goal of 5%.
Statistical Analysis 1: Comparison: Single Arm; The effectiveness endpoint for SMART MSP PAS is the proportion of the LV MSP Group with an Improved CCS. For this endpoint, those subjects in the LV MSP Group that become responders will be defined as having an Improved CCS. H0: Proportion of LV MSP Group subjects with Improved CCS from 6 Month Visit through 12 Month Visit ≤ 5%; Test type: Other — Even though fewer subjects (78) were available for the effectiveness endpoint analysis than originally planned (110), the study was still powered at approximately 90%; Proportion = 51.3, 95% CI 1-sided [lower limit 41.1]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from enrollment until the time the subject's participation ended. Subjects were considered to have completed the study after 12 months of follow up.
Description: Reportable adverse events included the following; All Serious Adverse Events, All Heart Failure and Cardiac related Adverse Events requiring IV or invasive therapy, including new onset of cardiac events, or worsening in severity or frequency of preexisting condition, All Adverse Device Effects, All Device Deficiencies, All Adverse Events relate to the protocol required testing, excluding PNS during lead testing ad Unanticipated Adverse Device Effects/Unanticipated Serious Adverse Device Effects.
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 19/584
Serious Adverse Events (participants affected / at risk) | 131/584
Other Adverse Events (participants affected / at risk) | 72/584
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=584)
Hematological (Blood and lymphatic system disorders) | 2 (2)
Atrial Fibrillation (AF) (Cardiac disorders) | 4 (5)
Atrial Tachycardia/Other SVT (eg AVRT, AVNRT, EAT) (Cardiac disorders) | 4 (4)
Cardiac arrest (Cardiac disorders) | 2 (2)
Cardiogenic shock (Cardiac disorders) | 3 (4)
Chest pain - Heart failure (Cardiac disorders) | 2 (2)
Dyspnea - Heart failure (Cardiac disorders) | 15 (22)
Gastrointestinal - Heart failure (Cardiac disorders) | 1 (1)
Heart failure symptoms - Unspecified (Eye disorders) | 8 (10)
Incessant VT/VT Storm (Cardiac disorders) | 1 (1)
Mitral regurgitation (Cardiac disorders) | 2 (2)
Multi-system failure - Heart failure (Cardiac disorders) | 1 (1)
Multiple Ventricular Arrhythmias (Cardiac disorders) | 1 (1)
Multiple heart failure symptoms (Cardiac disorders) | 22 (28)
Other - Heart failure patient condition- Cardiovascular (Cardiac disorders) | 4 (4)
Other - Patient condition - Cardiovascular (Cardiac disorders) | 1 (2)
Palpitations (Cardiac disorders) | 1 (1)
Pericardial effusion - Unrelated (non study) procedure or device (Cardiac disorders) | 1 (1)
Pulmonary edema - Heart failure (Cardiac disorders) | 3 (3)
Renal insufficiency/failure - Heart failure (Cardiac disorders) | 1 (1)
Valvular damage/Valvular insufficiency (Cardiac disorders) | 2 (2)
Ventricular Fibrillation (VF) (Cardiac disorders) | 1 (1)
Ventricular Tachycardia (VT)/Monomorphic VT (Cardiac disorders) | 8 (8)
Weight gain - Heart failure (Cardiac disorders) | 2 (2)
Atrial (Type 1) Flutter (Cardiac disorders) | 1 (1)
Gastrointestinal (Gastrointestinal disorders) | 12 (13)
Endocrine (Endocrine disorders) | 1 (1)
Chest Pain - Other (General disorders) | 5 (7)
Death (General disorders) | 2 (2)
Fatigue and Weakness (General disorders) | 3 (3)
HEENT (General disorders) | 2 (2)
Multi-System Failure (General disorders) | 2 (2)
Other-Patient Condition-Non-Cardiovascular (General disorders) | 1 (1)
Physical Trauma (General disorders) | 3 (3)
Syncope (General disorders) | 4 (4)
Fever and/or Virus (Infections and infestations) | 1 (1)
Infection (>30 days post-implant) - PG System - Subject related (Infections and infestations) | 4 (4)
Localized Infection (Infections and infestations) | 2 (2)
Systemic Infection (Infections and infestations) | 4 (4)
Hematoma - Pocket (<=30 days post-implant) (Injury, poisoning and procedural complications) | 3 (3)
Post-surgical infection (<=30 days post-implant) (Injury, poisoning and procedural complications) | 2 (2)
Seroma - Pocket (<=30 days post-implant) (Injury, poisoning and procedural complications) | 1 (1)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 3 (3)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5)
Neurological (Nervous system disorders) | 4 (5)
Dislodgement - LV (Product Issues) | 2 (2)
Dislodgement - RA (Product Issues) | 3 (4)
Dislodgement - RV (Product Issues) | 2 (2)
Erosion - PG System - Subject related (Product Issues) | 1 (1)
Inappropriate Tachy Therapy - SVT - PG System Therapy (Product Issues) | 1 (1)
Inappropriate tachy therapy - SVT - Defibrillation lead (Product Issues) | 3 (4)
Genitourinary (Renal and urinary disorders) | 7 (8)
Renal (Renal and urinary disorders) | 14 (16)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 10 (11)
Integumentary (Skin and subcutaneous tissue disorders) | 1 (1)
Cerebrovascular Accident (CVA) - unspecifed (Vascular disorders) | 2 (2)
Coronary Artery Disease (Vascular disorders) | 3 (3)
Hematoma - Unrelated (non study) procedure or device (Vascular disorders) | 1 (1)
Hypotension/Orthostatic Hypotension (Vascular disorders) | 1 (1)
Myocardial Infacrtion (Vascular disorders) | 5 (5)
Pseudoaneurysm with hematoma (Vascular disorders) | 1 (1)
Pulmonary Embolism (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=584)
Premature Atrial Contraction (PAC) (Cardiac disorders) | 1 (1)
Premature Ventricular Contractions (PVC) (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Ventricular Fibrillation (VF) (Cardiac disorders) | 1 (1)
Ventricular Tachycardia (VT)/Monomorphic VT (Cardiac disorders) | 2 (3)
Weight gain - Heart failure (Cardiac disorders) | 1 (1)
Gastrointestinal (Gastrointestinal disorders) | 2 (2)
Abnormal laboratory values (General disorders) | 1 (2)
Adverse reaction - Medication (General disorders) | 1 (1)
Chest pain - Other (General disorders) | 1 (1)
Dizziness (General disorders) | 1 (1)
Head, eyes, ears, nose, throat (HEENT) (General disorders) | 1 (1)
Multiple symptoms (General disorders) | 1 (1)
Other - Patient condition- Non-cardiovascular (General disorders) | 1 (1)
Physical trauma (General disorders) | 1 (1)
Localized Infection (Infections and infestations) | 1 (1)
Hematoma - Pocket (<=30 days post-implant) (Injury, poisoning and procedural complications) | 2 (2)
Post-surgical infection (<=30 days post-implant) (Injury, poisoning and procedural complications) | 2 (2)
Post-surgical wound discomfort/bruising/swelling (Injury, poisoning and procedural complications) | 2 (2)
Thromboembolic events (Injury, poisoning and procedural complications) | 1 (1)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 3 (3)
Dislodgment - RA (Product Issues) | 1 (1)
Elevated threshold - LV Lead (Product Issues) | 3 (3)
Extracardiac stimulation - LV Lead (Product Issues) | 21 (22)
Extracardiac stimulation - RV Lead (Product Issues) | 1 (1)
Inappropriate tachy therapy - NSR -Defibrillation lead (Product Issues) | 1 (1)
Inappropriate tachy therapy - SVT - Defibrillation lead (Product Issues) | 1 (1)
Pacemaker Mediated Tachycardia - PG System Therapy (Product Issues) | 8 (8)
Genitourinary (Renal and urinary disorders) | 1 (1)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Integumentary (Skin and subcutaneous tissue disorders) | 1 (1)
Arterial/venous thrombolytic event (Vascular disorders) | 1 (1)
Chest pain - Ischemic (Vascular disorders) | 1 (1)
Hypotension/Orthostatic Hypotension (Vascular disorders) | 1 (1)
Peripheral vascular disease (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Because the study was not designed to randomize subjects to conventional CRT or LV MSP, the potential incremental benefit of LV MSP cannot be quantified.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-15): https://cdn.clinicaltrials.gov/large-docs/36/NCT03257436/Prot_SAP_000.pdf